CLINICAL TRIAL: NCT03725995
Title: The Effectiveness of Topical Lidocaine in Relieving Pain Related To Intranasal Midazolam Sedation: A Randomized, Placebo-Controlled Clinical Trial
Brief Title: Using Intranasal Midazolam (INM) and Lidocaine for Uncooperative Children
Acronym: INM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Principal Investigator, Nabih Raslan, Principal Investigator, Tishreen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tishreen U- PediatricDentistry
Record Dates: First submitted 2018-10-21; First posted 2018-10-31 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Burning Nose
Keywords: midazolam; Lidocaine; Intranasal; Burning; Children
MeSH Terms: conditions — Paresthesia | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: blinded, randomized placebo-controlled trial, comparing three groups.
Who Masked: Participant, Investigator
Masking Description: The participant was blinded, the first assistant who explained the pain scale to the participants and asked him\her to record the score of pain associated with the drug administration was also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A (Midazolam) (Active Comparator): 21 children received 0.5 mg/kg intranasal medication (midazolam), with a maximum dose of 10 mg, via a spray of 0.2 ml per puff, administering the drug was alternated between the two nostrils of the child.
  Interventions: Drug: Midazolam
- B (Lidocaine-Midazolam) (Experimental): 21 children received a puff of lidocaine 2% in each nostril, after 60 seconds, they received 0.5 mg/kg intranasal medication (midazolam),administering the drug was alternated between the two nostrils of the child, with a maximum dose of 10 mg via a spray of 0.2 ml per puff.
  Interventions: Drug: Lidocaine-Midazolam
- C (Placebo) (Placebo Comparator): 21 children received intranasal medication (saline 9% as placebo), 0.5 mg/kg, with a maximum dose of 10 mg via a spray of 0.2 ml per puff,administering the drug was alternated between the two nostrils of the child.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midazolam — Patients received 0.5 mg/kg midazolam, with a maximum dose of 10 mg, Immediately following the administration, the child was asked to record the score of pain on the self reporting pain scale, WBFS.
  Other Names: A
  Arms: A (Midazolam)
Drug: Lidocaine-Midazolam — Patients received a puff of lidocaine 2% in each nostril, after 60 seconds, they received 0.5 mg/kg midazolam, with a maximum dose of 10 mg. , Immediately following the administration, the child was asked to record the score of pain on the self reporting pain scale, WBFS.
  Other Names: B
  Arms: B (Lidocaine-Midazolam)
Drug: Placebo — Patients received saline 9% (placebo), 0.5 mg/kg, with a maximum dose of 10 mg, Immediately following the administration, the child was asked to record the score of pain on the self reporting pain scale, WBFS.
  Other Names: C
  Arms: C (Placebo)

SUMMARY:
Aims: The objective of the current study was to evaluate the effectiveness of topical lidocaine in relieving pain related to INM administration.

Design: This was a blinded, randomized placebo-controlled trial. Sixty-three uncooperative children, aged 4 - 11.

DETAILED DESCRIPTION:
Background and Aims: The use of intranasal midazolam (INM) has been commonly associated with a burning sensation of the nasal mucosa. However, despite its significance, this subject has received little adequate research focus. The objective of the current study was to evaluate the effectiveness of topical lidocaine in relieving pain related to INM administration.

Design: This was a blinded, randomized placebo-controlled trial. Sixty-three uncooperative children, aged 4 - 11, were randomly assigned to one of three groups to receive the drug nasally via a pre-calibrated spray as per the following assignments:

A: received 0.5 mg/kg midazolam, B: received lidocaine 2% prior to 0.5 mg/kg midazolam.

C: received saline 9% (placebo), 0.5mg/kg. Children were asked to record the degree of pain using Wong-Baker-Faces- (WBFS) Scale.

ELIGIBILITY:
Inclusion Criteria:

* uncooperative children scored 1 or 2 on Frankle Scale.
* had no medical history of neurological or cognitive alterations.
* No facial deformities.
* ASA Classification I.
* requiring dental treatment under local anesthesia.

Exclusion Criteria:

* known allergy to midazolam or any other benzodiazepines.
* upper respiratory tract infection with nasal discharge.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Scores on the Wong Baker Faces Scale for pain assessment when administering midazolam alone, saline or midazolam premidicated with lidocaine . | one to five minutes following the administration.
  The use of intranasal midazolam is associated with a burning sensation of the nasal mucosa, the pain was assessed using a self report pain scale Wong Baker Faces Scale, the degree of pain is determined by choosing a score of (0-2-4-6-8-10) (minimum score 0, means no pain, maximum score 10, means the drug hurts worst, higher scores are worse) the scores were reported by children received intranasal midazolam alone, intranasal midazolam preceded by intranasal lidocaine or intranasal saline (placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Raslan, Dr., Study Chair — Tishreen University; Walaa Khalil, Dr., Principal Investigator — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Undecided
up to date, there is no decision about IPD sharing.

REFERENCES:
- [Result] Smith D, Cheek H, Denson B, Pruitt CM. Lidocaine Pretreatment Reduces the Discomfort of Intranasal Midazolam Administration: A Randomized, Double-blind, Placebo-controlled Trial. Acad Emerg Med. 2017 Feb;24(2):161-167. doi: 10.1111/acem.13115. Epub 2017 Jan 30. PMID 27739142